CLINICAL TRIAL: NCT01304563
Title: Safety and Efficacy of Dose Sparing Intradermal 2010/2011 Trivalent Influenza Vaccination With the Novel Microneedle Delivery Device
Brief Title: 2010/2011 Trivalent Influenza Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Dr Ivan FN Hung, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKU-2010-149
Record Dates: First submitted 2011-02-23; First posted 2011-02-25 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- IM15 (Active Comparator): 15 mcg TIV 2010/2011 influenza vaccine delivered via intramuscular injection (control)
  Interventions: Biological: TIV 2010/2011 influenza vaccine
- ID1 (Active Comparator): Low dose TIV 2010/2011 influenza vaccine delivered via intradermal injection (MicronJet)
  Interventions: Biological: TIV 2010/2011 influenza vaccine
- ID2 (Active Comparator): Higher low dose TIV 2010/2011 influenza vaccine delivered via intradermal injection (MicronJet)
  Interventions: Biological: TIV 2010/2011 influenza vaccine
- INT (Active Comparator): Low dose TIV 2010/2011 influenza vaccine delivered via a short needle intradermal device
  Interventions: Biological: INT

INTERVENTIONS:
Biological: TIV 2010/2011 influenza vaccine — TIV 2010/2011 influenza vaccine Intramuscular: 15 mcg TIV 2010/2011 vaccine x 1: Control
  Arms: IM15
Biological: TIV 2010/2011 influenza vaccine — Low dose TIV 2010/2011 influenza vaccine delivered via intradermal injection x 1: Experimental
  Arms: ID1
Biological: TIV 2010/2011 influenza vaccine — Higher lower dose TIV 2010/2011 influenza vaccine delivered via intradermal injection x 1: Experimental
  Arms: ID2
Biological: INT — Low dose TIV 2010/2011 influenza vaccine delivered via a short needle intradermal device x 1: Experimental
  Arms: INT

SUMMARY:
Intradermal influenza vaccination may result in better efficacy when compare to intramuscular vaccination.

DETAILED DESCRIPTION:
This is a prospective, randomized, single centre trial in the Queen Mary Hospital. We aim to recruit 400 subjects [with a minimum of 50 subjects per group] who would be qualified for the Hospital Authority (HA)/ Centre for Health Protection (CHP) Mass Vaccination Program for 2010/2011 TIV. These patients include all elderly at the age of 65 or above and all adult patients at the age of 21 or above with chronic illness (or healthcare workers). Subjects will be randomly assigned into 4 groups: Group 1 (ID1) to receive a single low-dose intradermal injection of 2010/2011 TIV, with a microneedle device. Group 2 (ID2) to receive a single higher low-dose intradermal injection of 2010/2011 TIV with a microneedle device. Group 3 (IM15) to receive a single full-dose (15ug) standard 2010/2011 TIV delivered intramuscularly by conventional needle. Group 4 (INT) to receive a single low-dose intradermal injection of 2010/2011 TIV, with Intanza® needle. The 2010/2011 TIV used will be Fluzone®, Sanofi-Pasteur for group 3 and Intanza®, Sanofi-Pasteur for group 1,2 and 4.

ELIGIBILITY:
Inclusion Criteria:

* All participants qualified for the HA/ CHP Mass Vaccination Program for TIV 2010/2011 seasonal influenza as stated above: including all elderly at the age of 65 or above and all adult patients at the age of 21 or above that are either healthcare workers or that have a chronic illness including hypertension, diabetes mellitus, ischemic heart disease, cerebrovascular disease, thyroid disease and chronic renal failure.
* All patients give written informed consent.
* Subjects must be available to complete the study and comply with study procedures.

Exclusion Criteria:

* Clinically significant immune-related diseases, significant recent co-morbidities and pregnant volunteers.
* History or any illness that might interfere with the results of the study or pose additional risk to the subjects due to participation in the study
* Have a known allergy to eggs or other components of the Study Vaccines (including gelatin, formaldehyde, octoxinol, thimerosal, and chicken protein), or history of any anaphylaxis, serious vaccine reactions, to any excipients.
* Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months.
* Have an active neoplastic disease or a history of any hematologic malignancy.
* Have known active human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C infection or autoimmune hepatitis and cirrhosis.
* History of progressive or severe neurological disorders or Guillain-Barré Syndrome.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
seroconversion rate | day 21
  Seroconversion rate (percentage of subjects with a fourfold increase in antibody titres, providing a minimal post vacination titre of 1:40) on day 21 by TIV 2010/2011 hemagglutination inhibition (HI) between the ID and IM groups

SECONDARY OUTCOMES:
Adverse events | 30 minutes post vaccination
  Adverse events secondary to vaccination with different devices
Seroprotection rate | Day 21
  percentage of subjects with a post vaccination titre of at least 1:40

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong, China